CLINICAL TRIAL: NCT04841980
Title: Rifaximin Therapy Versus Low FODMAP Diet In Irritable Bowel Syndrome: A Randomised Controlled Trial
Brief Title: Rifaximin Therapy vs Low FODMAP Diet In IBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Chuah Kee Huat, Medical Lecturer and Clinical Specialist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021001
Record Dates: First submitted 2021-01-21; First posted 2021-04-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth
Keywords: Rifaximin; low FODMAP diet; IBS; SIBO
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Rifaximin; FODMAP Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics (Active Comparator)
  Interventions: Drug: Rifaximin
- Dietary based therapy (Active Comparator)
  Interventions: Other: Low FODMAP diet

INTERVENTIONS:
Drug: Rifaximin — Administration route: PO Rifaximin 400mg TDS for 2 weeks
  Arms: Antibiotics
Other: Low FODMAP diet — Low FODMAP diet under dietitian guidance for 4 weeks
  Arms: Dietary based therapy

SUMMARY:
Functional gastrointestinal disorders (FGIDs) are common and from the most recent global epidemiology study, an estimated 40% of the world population suffer from the condition. FGIDs cause significant morbidity to patients, despite not influencing mortality. IBS is among the most important functional gastrointestinal disorder with an estimated 3.8 to 9.2 % of the general population worldwide were affected by this disorder.

Rifaximin (gut specific antibiotic) and low FODMAP diet (dietary based therapy) were proven to be effective in treating irritable bowel syndrome (IBS), however there was no head-to-head study comparing both treatments. This study will help doctors to understand the efficacy of different IBS/SIBO treatments. With the evaluation of factors that can predict treatment response, doctor could potentially treat IBS and SIBO more effectively in future.

The purpose of the study is to compare the clinical symptoms and psychological improvement in patients with irritable bowel syndrome (IBS) after treatment with Rifaximin versus treatment with low FODMAP diet. The factors that is associated with treatment response will also be evaluated. In IBS patients with small intestinal bacterial overgrowth (SIBO), eradication rate of SIBO will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Irritable bowel syndrome using Rome III diagnostic criteria with Abdominal Pain/ Discomfort Intensity of weekly average of worst abdominal pain/ discomfort in past 24 hours score of ≥ 3.0 on a 0 to 10 point scale AND Stool Consistency of at least 2 days per week with at least one stool that has a consistency of Type 6 or Type 7 BSS or <3 CSBM per week
2. Subject who can provide written informed consent and willingness to comply with the requirement of the protocol
3. Able to communicate in English, Malay, or Mandarin languages

Exclusion Criteria:

1. Patients with known hypersensitivity or contraindication to Rifaximin
2. Pregnant / breastfeeding women
3. Patients who are on probiotics for the past 1 month
4. Presence of family history of GI malignancy or alarm features suggested malignancy - e.g. Unintentional weight loss (≥ 10% of body weight in recent 6 months), GI bleeding
5. History of gastrointestinal (GI) malignancy
6. Patients with any hepatobiliary or pancreatic diseases
7. Patients with severe depression, anxiety, or other psychological disorder
8. Patients with any terminal disease
9. Other conditions determined by the investigator to be inappropriate for this clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with adequate relief of composite of abdominal symptom (pain/discomfort) and stool symptom (frequency/ consistency) after treatment. | 4 weeks
  Adequate relief was defined as self-reported relief of both symptoms (abdominal symptom and stool symptom) at least in week 2 or 4. (Subjects will be provided with self-reported questionnaires for week 2 and 4).
  For IBS-D, relief was defined as a decrease of at least 30% from baseline in weekly mean ratings of IBS-related abdominal pain or discomfort and a weekly decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
  For IBS-C, relief was defined as a decrease of at least 30% from baseline in weekly mean ratings of IBS-related abdominal pain or discomfort and an increase of 1 or more complete spontaneous bowel movement (CSBM) per week compared with baseline.
  For IBS-M, relief was defined as fulfilled both IBS-D and IBS-C symptom relief criteria.

SECONDARY OUTCOMES:
Proportion of patients who had relief was determined from the patients' weekly assessments of global IBS symptoms, bloating, abdominal pain/ discomfort, and stool consistency/ frequency after treatment with Rifaximin or low FODMAP diet | 4 weeks
  Rated on a 5-point scale: 2 = Significantly Relieved, 1 = Moderately Relieved, 0 = Unchanged, -1 = Moderately Worse, and -2 = Significantly Worse for at least 50% of the days in a week.
  Relief was defined as a score of either 2 (Significantly Relieved) or 1 (Moderately Relieved).
Symptom severity score improvement | 4 weeks
  The symptom severity was assessed by the IBS-symptom severity (IBS-SS) score from baseline to 4 weeks after initiation of treatment. Total scores ranging from 0 to 500
Proportion of patients with SIBO who had eradication of SIBO after treatment | 6 weeks
  as measured by glucose hydrogen breath test
Assessment of factors that were associated with treatment response | 6 weeks
  Baseline characteristic (age, gender, ethnicity), IBS subtype (IBS-D, IBS-C IBS-mixed), and SIBO status (positive or negative) of patients who responded to treatment (based on primary outcome) will be compared to non-responder
Change in Health-Related Quality of Life (HRQOL) score | 4 weeks
  HRQOL will be assessed using EuroQol-5D (EQ-5D) instrument. Overall utility score (as mean value) was calculated with a range score from 0 (worst health scenario) to a maximum of 1.0 (best health scenario).

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Huat Chuah, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuah KH, Loo QY, Loh AJC, Leong JY, Chan WL, Khoo XH, Wong KL, Panirsheeluam S, Natarajan V, Ng AK, Abdul Majid H, Mahadeva S. Clinical Trial: Rifaximin Versus Low FODMAP Diet in Irritable Bowel Syndrome. Aliment Pharmacol Ther. 2026 Jan;63(2):210-221. doi: 10.1111/apt.70420. Epub 2025 Oct 16. PMID 41098003